CLINICAL TRIAL: NCT05433324
Title: "Long COVID-19" on the Human Brain
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 139/2021
Record Dates: First submitted 2022-06-23; First posted 2022-06-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Long Covid; Post Acute Sequelae of COVID-19
Keywords: Magnetic resonance imaging; Positron emission tomography
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and nasopharyngeal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: Persons previously infected with COVID-19 experiencing CNS-PASC within 6 months of recovery
  Interventions: Other: MRI and PET Scans
- Group B: Persons previously infected with COVID-19 without CNS-PASC symptoms within 6 months of recovery
  Interventions: Other: MRI and PET Scans
- Group C: A control group of persons not previously infected with COVID-19.
  Interventions: Other: MRI and PET Scans

INTERVENTIONS:
Other: MRI and PET Scans — All groups will undergo cognitive tests and brain imaging scans (MRI & PET)

SUMMARY:
Over one million Canadians have been infected by COVID-19. Many people who have been infected by COVID-19 experience negative mental symptoms, such as "brain fog" and fatigue. For many of these people, they continue to feel these negative mental symptoms even after recovering from COVID-19. However, scientists still do not know how COVID-19 harms the human brain and causes these mental problems. Our goal is to use advanced brain imaging to determine whether people who have been infected with COVID-19 show damage in their brain. We hope that this information will help doctors determine what treatments should be provided to help people who are suffering from continuing mental problems after being infected with COVID-19.

DETAILED DESCRIPTION:
This is a cross-sectional study composed of three participant groups. 1) persons previously infected with COVID-19 experiencing CNS-PASC (central nervous system Post-Acute Sequelae of COVID-19) within 6 months of recovery, 2) persons previously infected with COVID-19 without CNS-PASC symptoms within 6 months of recovery, and 3) a control group of persons not previously infected with COVID-19. Groups will be as similar as possible for age and substance use. This study will examine synaptic vesicular density (henceforth, synaptic density), as measured with positron emission tomography (PET), and neuroinflammation markers, as measured with Magnetic resonance imaging (MRI), as well as clinical, cognitive, and peripheral biomarkers between the groups.

Participants that meet the inclusion and exclusion criteria at the initial screening visit (Visit 1) and provide written consent will be enrolled into the study. Participants will undergo PET scans with the novel PET tracer [18F]SDM-8 to quantify synaptic density levels. MRI scans will be collected, and clinical assessments will be completed at the same time. Each participant will participate in four study visits at defined time points over the course of their enrolment, including the initial participant screening visit (Visit 1). Brain imaging scans and PASC/cognitive assessments will occur at visits 2 and 3, followed by a subsequent PASC/cognitive assessment follow-up at visit 4, occurring 2-3 months after Visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Persons of all races, ethnicities, genders, and sex.
2. 18 years of age or older.
3. Fully vaccinated for COVID-19 with authorized vaccines in Canada.

Participants in COVID-19 groups (Group A and B) will have the following additional inclusion criteria:

1. Previously infected with mild-moderate COVID-19 (i.e., out-patients never hospitalized for COVID-19), as confirmed by review of clinical history.
2. Not currently infected with SARS-COV-2, as confirmed by COVID-19 Rapid Antigen Test (RAT).

Additionally, participants enrolled as part of the CNS-PASC group (Group A), must also:

1. Currently experience CNS-PASC symptoms, not present prior to infection, as confirmed by the "Long COVID-19 Symptom Assessment" scale.

Exclusion Criteria:

Participants will be excluded if they meet ANY of the criteria listed below:

1. Unstable medical conditions and/or active uncontrolled autoimmune or inflammatory conditions.
2. Neurological conditions and/or concussion present prior to COVID-19 infection.
3. Substance abuse disorder (except caffeine, nicotine, and cannabis/marijuana) within 6 months of entering the study, as determined by the Structured Clinical Interview (37)
4. Positive urine drug screen for drugs of abuse at the screening visit (except for cannabis/marijuana).
5. Pregnancy (Note: Females up to age 65 must have negative urine pregnancy test at screening), or breastfeeding.
6. Score <32 on the Wide Range Achievement Test-III.
7. Receiving treatment with medications such as levetiracetam that blocks SV2a binding.
8. Pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or any other conditions that would preclude the MRI scan.
9. Body size/weight above the limits for PET and MRI scanners.
10. Exceeding allowed annual radiation exposure levels for research scans of 20 mSv in the past 12 months as outlined by our PET Centre guidelines.
11. Having completed multiple PET scans in the past, such that participation in this study would cause participant to exceed lifetime limit (8 PET scans).
12. Currently receiving active treatment for cancer.
13. Claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with or without prior infection with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Synaptic Density (PET Scan) | At baseline
  [18F]SDM-8's regional binding potential non-displaceable (BPND) will be calculated using the simplified reference tissue model (SRTM) (31) using as reference the centrum semiovale (32). The PET data will be analyzed using both a priori regions of interest and exploratory whole-brain voxel-based analysis method.
Presence and Severity of CNS and PASC Symptoms | At screening, baseline and at 3-month follow-up
  A Likert-type scale of the most common COVID-19 sequela symptoms will be employed. The "Long COVID-19 Symptom Assessment" self-report consists of 46 common COVID-19 sequela symptoms, both neurological and non-neurological.

SECONDARY OUTCOMES:
Changes in Quality of Life | At baseline and at 3-month follow-up
  The World Health Organization Disability Assessment Schedule (WHODAS 2.0) will be administrated. The WHODAS 2.0 is a short, easily administered test that takes approximately 5-20 minutes to complete. It covers 6 domains of function to assess a person's quality of life which include cognition, mobility, self-care, getting along, life activities and participation.
Cognitive, Emotional, Motor and Sensation Measures | At baseline and at 3-month follow-up
  Assessment of neurological and behavioural function will be done using the National Institute of Health (NIH) Toolbox (www.nihtoolbox.org). The measures in the toolbox are administered in two hours and have been validated for the assessment of longitudinal epidemiologic outcomes.
Biomarker Measures | At screening, baseline and at 3-month follow-up
  COVID-19 Humoral Status, CNS Humoral Autoreactivities in Tissue Microarrays, Biobanking of Live PBMC, COVID-19-specific T Cell Cytokine Response, Mucosal immune response, Metabolic Markers

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Graff, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — https://www.camh.ca/en/science-and-research